CLINICAL TRIAL: NCT04094519
Title: A Phase 1 Open-label Study to Evaluate the Effect of Multiple Doses of Enzalutamide on the Pharmacokinetics of Substrates of P-glycoprotein (Digoxin) and Breast Cancer Resistant Protein (Rosuvastatin) in Male Subjects With Prostate Cancer
Brief Title: A Study to Evaluate the Effect of Multiple Doses of Enzalutamide on the Pharmacokinetics of Substrates of P-glycoprotein (Digoxin) and Breast Cancer Resistant Protein (Rosuvastatin) in Male Subjects With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0018
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: ASP9785; enzalutamide; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- digoxin plus rosuvastatin and enzalutamide (Experimental): Participants will receive a single oral dose cocktail containing 0.25 mg digoxin and 10 mg rosuvastatin on Day 1 and 64. A single oral dose of placebo to match enzalutamide will be given on Day 1 and 160 mg enzalutamide once daily on Days 8 through 71.
  Interventions: Drug: enzalutamide; Drug: enzalutamide Placebo; Drug: digoxin; Drug: rosuvastatin

INTERVENTIONS:
Drug: enzalutamide — oral
  Other Names: ASP9785
Drug: enzalutamide Placebo — oral
Drug: digoxin — oral
Drug: rosuvastatin — oral

SUMMARY:
The primary purpose of this study is to determine the effect of multiple once daily administrations of enzalutamide on the pharmacokinetics of a single dose of digoxin (P-glycoprotein (P-gp) substrate) and rosuvastatin (breast cancer resistant protein (BCRP) substrate) in participants with prostate cancer.

This study will also evaluate the safety and tolerability of multiple once daily administrations of enzalutamide alone and in combination with a single dose of digoxin (P-gp substrate) and rosuvastatin (BCRP substrate) in participants with prostate cancer, as well, assess the pharmacokinetics of enzalutamide and its active metabolite.

DETAILED DESCRIPTION:
Eligible participants will be admitted to the clinical unit on day -1. Participants may be discharged from the clinical unit on day 2 on the condition that all required assessments have been performed and that there are no medical reasons for a longer stay in the clinical unit and participants are able and willing to return to the clinical unit on days 3 to 8 for daily pharmacokinetic sampling. Or, participants may choose to remain in the clinical unit up to the 168 hour postdose (day 8) pharmacokinetic sample collection.

Participants will return to the clinical unit on day 35 for an ambulant visit and will be admitted to the clinical unit on day 63. Participants may be discharged from the clinical unit on day 65 on the condition that all required assessments have been performed and that there are no medical reasons for a longer stay in the clinical unit and participants are able and willing to return to the clinical unit on days 66 to 71 for daily pharmacokinetic sampling. Or, participants may choose to remain in the clinical unit up to the 168 hour postdose (day 71) pharmacokinetic sample collection.

From day 72 onwards, participants experiencing clinical benefit (determined by the investigator in consultation with the physician responsible for treating the participants' prostate cancer) may roll over into an open label, single arm extension study. Only participants who will be enrolled into the extension study will continue to receive enzalutamide until any discontinuation criterion occurs per the extension study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation, signet cell or small cell histology.
* Subject has a serum testosterone level < 1.7 nmol/L (50 ng/dL) during the screening period if under androgen deprivation therapy (ADT).
* Subject has newly diagnosed metastatic prostate cancer or progressive disease on ADT confirmed by prostate-specific antigen (PSA) or imaging. Disease progression at screening is defined as 1 or more of the following 3 criteria:

  * PSA progression defined by a minimum of 2 rising PSA levels with an interval of ≥ 1 week between each determination. At least 1 PSA value within the 3 months leading up to the screening period should be ≥ 2μg/L (2 ng/mL).
  * Soft tissue disease progression defined by the Response Evaluation Criteria in Solid Tumors, version 1.1 for soft tissue disease.
  * Bone disease progression defined by 2 or more new lesions on a bone scan.
* Subject is able to swallow enzalutamide capsules and comply with study requirements.
* Subject has an Eastern Cooperative Oncology Group performance status of 0 to 2.
* Subject with a female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 3 months after final investigational product (IP) administration.
* Subject must not donate sperm during the treatment period and for 3 months after final IP administration.
* Subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 3 months after final IP administration.
* Subject has a body mass index range of 18.5 to 35.0 kg/m2 inclusive. The subject weighs at least 50 kg at screening.
* Subject has an estimated life expectancy of at least 6 months.
* Subject agrees not to participate in another interventional study while receiving IP treatment in the present study/participating in the present study.

Exclusion Criteria:

* Subject has any condition, which makes the subject unsuitable for study participation or is not likely to complete the study for any reason.
* Subject has known metastases in the liver or any hepatic disorder that could affect drug metabolism deemed clinically significant.
* Subject is self-reported as Asian.
* Subject has known or suspected brain metastasis or active leptomeningeal disease.
* Subject has a history of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma, brain arteriovenous malformation).
* Subject has a history of loss of consciousness or transient ischemic attack within 12 months of day 1.
* Subject has clinical signs suggestive of high or imminent risks for pathological fracture, spinal cord compression and/or cauda equine syndrome.
* Subject has clinically significant cardiovascular disease including the following:

  * Myocardial infarction within 6 months before screening
  * Unstable angina within 3 months before screening
  * New York Heart Association class III or IV congestive heart failure or a history of New York Heart Association class III or IV congestive heart failure, unless a screening echocardiogram or multigated acquisition scan performed within 3 months before screening demonstrates a left ventricular ejection fraction ≥ 45%
  * History of clinically significant ventricular arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes)
  * History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place
  * Hypotension as indicated by systolic blood pressure < 86 mm Hg at screening
  * Bradycardia as indicated by a heart rate of ≤ 45 beats per minute on the screening electrocardiogram (ECG)
  * Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg at screening
* Subject has previously received treatment with enzalutamide.
* Subject has undergone major surgery within 4 weeks prior to day 1.
* Subject has a known hypersensitivity reaction to enzalutamide, digoxin, rosuvastatin, contrast agents or any of the components of the formulations used.
* Subject has an absolute neutrophil count < 1500/μL, platelet count < 100000/μL and hemoglobin < 6.2 mmol/L (9 g/dL) during the screening period.
* Subject has received any growth factors or blood transfusions within 7 days prior to the hematologic laboratory values obtained during the screening period.
* Subject has a total bilirubin (TBL) > 1.5 times the upper limit of normal (ULN) (except for subjects with documented Gilbert's disease), alanine aminotransferase (ALT) > 2.5 times the ULN or aspartate aminotransferase (AST) > 2.5 times the ULN during the screening period. Subject with alkaline phosphatase (ALP) > 3 times ULN will be excluded, unless deemed to be related to bone metastasis, rather than liver disease, and after discussion with the sponsor's medical monitor.
* Subject has an albumin < 30 g/L (3.0 g/dL) or creatinine > 177 μmol/L (> 2 mg/dL) during the screening period.
* Subject has clinical signs and symptoms of hereditary or acquired coagulation disorders within 6 months prior to enrollment (day 1 visit).
* Subject has a history of another invasive cancer within 3 years before screening, with the exception of fully treated cancers with a remote probability of recurrence. The medical monitor and investigator must agree that the possibility of recurrence is remote.
* Subject received treatment with chemotherapy within 4 weeks prior to enrollment (day 1) or plans to initiate treatment with chemotherapy during the study.
* Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 28 days or 5 half-lives, whichever is longer, prior to the initiation of screening.
* Subject has a gastrointestinal disorder affecting absorption.
* Subject uses concomitant medications that are inducers or inhibitors of P-gp and/or BCRP or strong CYP2C8 inhibitors or strong CYP3A4 inducers.
* Subject uses digoxin or rosuvastatin or concomitant medications that are contraindicated with digoxin or rosuvastatin.
* Subject has any history or evidence of any clinically significant gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease.
* Subject has used drugs of abuse (if not medically indicated) within 3 months prior to admission to the clinical unit.
* Subject has a history of consuming > 21 units of alcohol per week within 3 months prior to day -1 (note: 1 unit = 10 g pure alcohol, 250 mL of beer [5%], 35 mL of spirits [35%] or 100 mL of wine [12%]) or the subject tests positive for alcohol at screening or on day -1.
* Subject has known active hepatitis B (hepatitis B surface antigen [HBsAg] reactive, associated with positive anti-hepatitis B core and detectable hepatitis B virus DNA), active hepatitis C (hepatitis C virus [HCV] RNA [qualitative] is detected) or active viral hepatitis A (immunoglobulin M).
* Subject has a positive human immunodeficiency virus type 1 and/or type 2 at screening.
* Subject is an employee of Astellas, the study-related contract research organizations (CRO) or the clinical unit.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-12-27 (Actual); Study Completion 2020-12-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of Digoxin in combination with rosuvastatin in plasma: maximum concentration (Cmax) | Up to Day 71
  Cmax will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of Digoxin in combination with rosuvastatin in plasma: area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast) | Up to Day 71
  AUClast will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of Digoxin in combination with rosuvastatin in plasma: area under the concentration time curve from the time of dosing extrapolated to time infinity (AUCinf) | Up to Day 71
  AUCinf will be recorded from the pharmacokinetic (PK) plasma samples collected.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Day 101
  Adverse events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA).
  An AE is any untoward medical occurrence in a participant administered an Investigational Product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of IP whether or not considered related to the IP.
  An AE is considered "serious" if the event: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly or birth defect; requires inpatient hospitalization (except for planned procedures)or leads to prolongation of hospitalization (except if prolongation of planned hospitalization is not caused by an AE); or other medically important events.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to Day 101
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and /or adverse events (AEs) | Up to Day 101
  Number of participants with potentially clinically significant vital sign values.
Number of participants with routine 12-lead electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to Day 101
  Number of participants with potentially clinically significant ECG values.
Pharmacokinetics (PK) of enzalutamide and its metabolite (N-desmethyl) in plasma: maximum concentration (Cmax) | Up to Day 71
  Cmax will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of enzalutamide and its metabolite (N-desmethyl) in plasma: area under the concentration-time curve during a dosing interval, where tau (τ) is the length of the dosing interval (AUCtau) | Up to Day 71
  AUCtau will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of enzalutamide and its metabolite (N-desmethyl) in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to Day 71
  Ctrough will be recorded from the pharmacokinetic (PK) plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Site MD37301, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Poondru S, Ghicavii V, Khosravan R, Manchandani P, Heo N, Moy S, Wojtkowski T, Patton M, Haas GP. Effect of enzalutamide on PK of P-gp and BCRP substrates in cancer patients: CYP450 induction may not always predict overall effect on transporters. Clin Transl Sci. 2022 May;15(5):1131-1142. doi: 10.1111/cts.13229. Epub 2022 Feb 4. PMID 35118821
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/?pid=9785-CL-0018
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14668&tenant=MT_AST_9011